CLINICAL TRIAL: NCT03060759
Title: Light Therapy as Treatment for Fatigue in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Farrah Mateen, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P002696
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Relapsing-Remitting Multiple Sclerosis; Fatigue; Light Therapy
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light Therapy-Spectrum 1 (Active Comparator): Light from 'active' spectrum
  Interventions: Device: Light Therapy box
- Light Therapy-Spectrum 2 (Placebo Comparator): Light from 'placebo' spectrum
  Interventions: Device: Light Therapy box

INTERVENTIONS:
Device: Light Therapy box — The light box used for LT (SunRay by The Sunbox Company, Gaithersburg, Maryland, USA) is approximately 15.5" tall x 23" wide x 3.25" deep and is designed to stand on a desk or tabletop. It can be used both in the home or office. The light is delivered at a downward angle to maximize the effectiveness. The box runs on 124 watts and contains full spectrum 5000k 10,000 lux bulbs.

SUMMARY:
This prospective study will randomize 1:1 people living with multiple sclerosis-associated fatigue to one of two spectra of light therapy. Each participant will be asked to use the light box twice daily at home or at the workplace at preset hours during the day for a total of four weeks. Participants will be asked to record their fatigue on standard measurement scales before, during, and after the use of the light therapy box. The investigators anticipate a reduction in self-reported fatigue following the use of the light box therapy of a particular spectrum of light among people living with multiple sclerosis.

DETAILED DESCRIPTION:
Study Protocol:

Eligible participants will be consented and randomized 1:1 to (a) white LT (10,000 lux), or (b) dim red LT (<300 lux). Participants will be informed that this study will examine the effect of two different light spectra on fatigue. The following assessments will be administered by the study principal investigator at the baseline visit: (1) the Kurtzke Extended Disability Status Scale (EDSS), (2) FSS, (3) Beck Depression Inventory II (BDI), (4) Pittsburgh Sleep Quality Index (PSQI), (5) Berlin questionnaire for obstructive sleep apnea, (6) Epworth Sleepiness Scale. A two-week sleep diary will be collected before enrollment in order to screen for significant behavioral insufficient sleep or circadian rhythm disorders. The light box used for LT is designed to stand on a desk or tabletop. It can be used in the home or office. The light is delivered at a downward angle to maximize the effectiveness. The box runs on 124 watts and contains full spectrum 5000k 10,000 lux bulbs. Bright light treatment requires at least 2,500 lux to be effective.

Data Collection:

The study period will include a two-week baseline period, a four-week treatment period, and a four-week follow up period. Throughout the study period, participants will record their fatigue using the Visual Analogue Fatigue Scale (VAFS) four times daily, starting after waking up, and every four hours thereafter. The VAFS is a simple, validated 10-point scale ranging from 1 to 10 in which participants can report their fatigue as a snapshot at that particular moment. Data collection will occur by participants in self-report fashion. A FSS score will be collected at enrollment as well as at the end of the four week treatment period and the end of the four week follow-up period. There will be three visits with a principal investigators (PI), including the baseline visit described above, a visit with the PI at the end of the treatment period in which participants will report a FSS and discuss their experiences with LT, and a third follow-up visit at the end of the four-week follow up period for a final FSS. At this last visit they will be queried on whether they believe the intervention had any effect on their fatigue and whether they believe the alternative therapy (white light or dim red light) would have been more or less beneficial. Additionally participants will be asked to keep a LT log in which they will record daily LT exposure and associated side effects.

Statistical Analysis:

The primary outcome measure is the change in the average FSS after the four-week study period in the bright light "active" vs. dim light "control" groups. There are no reports on FSS in response to bright LT in pMS. Using the conventional values of α=0.05 and β=0.80 for 2-tailed tests of probability with equally sized groups: a difference in 10 points on FSS between groups requires 18 people per study arm; a difference in 8 points requires 28 people per group. If power is reduced to 70%, the sample sizes are 22 and 14 for 8-point and 10-point differences. First, the investigators will compare the mean change in FSS scores, from baseline to after completion of LT, in an intention to treat analysis. The secondary outcome measure will be a change in the global VAFS scores after light therapy in both groups. Frequencies will be used to describe baseline characteristics across treatment arms. X2 statistics or Fisher's exact test will be used to compare the differences between groups. VAFS will be evaluated using a mixed-effects model which accounts for correlation between repeated measurements. Participant logbooks will be used to generate summary statistics and graphically display fatigue patterns throughout the day. Logbooks will also qualitatively assess the safety and tolerability of LT.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing remitting Multiple Sclerosis based on the McDonald Criteria (2010)
* Over 18 years old
* Presence of fatigue defined as FSS over 36

Exclusion Criteria:

* A change in an anti-depressant up to 4 weeks prior to study screening
* A change in fatigue medication regime or MS disease modifying therapy up to 4 weeks prior to study screening
* Shift work
* Use of photosensitizing medication
* Presence of eye trauma or acute optic neuritis within the preceding 3 months
* History of traumatic brain injury
* Probable (untreated) sleep apnea based on Berlin questionnaire
* Significant anemia
* History of mania
* MS relapse in the preceding four weeks
* Current pregnancy
* Known light sensitivity
* Other complicating illness preventing study completion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Light Therapy-Spectrum 1 | Light Therapy-Spectrum 2
Started | 20 | 15
Completed | 15 | 12
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Light Therapy-Spectrum 1 | Light Therapy-Spectrum 2 | Total
Number analyzed (Participants) | 20 | 15 | 35
Age, Categorical [Count of Participants; unit: Participants] — Population: Row population is equal to overall population.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 20 | 15 | 35
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 47.2 [32 to 64] | 41.9 [25 to 60] | 44.9 [25 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 18 | 10 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 20 | 15 | 35
Years since first diagnosis [Mean (Full Range); unit: years] | 12.39 [1 to 30] | 8.93 [2 to 20] | 10.9 [1 to 30]
Expanded Disability Status Scale Score [Mean (Full Range); unit: units on a scale] — Scale of disability in MS. Range: 0 (normal neurological exam) to 10 (death due to MS). Lower scores indicate less disability.
  units on a scale | 3.1 [1 to 6] | 3.1 [1 to 6.5] | 3.1 [1 to 6.5]
Type of Multiple Sclerosis [Count of Participants; unit: Participants]
  Relapsing-remitting MS | 20 | 15 | 35
  Primary Progressive MS | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Fatigue Severity Scale (FSS) Score
Description: Measure of general level of fatigue. Range: 9 to 63. Lower scores indicate less reported fatigue.
Time Frame: 4 weeks
Population: 4 participants were withdrawn from the study before providing outcome data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Light Therapy-Spectrum 1 | Light Therapy-Spectrum 2
Number analyzed (Participants) | 17 | 14
score on a scale | 45.824 (11.8) | 46.714 (10.2)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 4 weeks of light therapy, with collection at 2 and 4 weeks after starting light therapy.
Description: 4 participants were withdrawn from the study prior to collection of adverse event data.
Arm/Group | Light Therapy-Spectrum 1 | Light Therapy-Spectrum 2
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 15/17 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Light Therapy-Spectrum 1 (N=17) | Light Therapy-Spectrum 2 (N=14)
Headache (Nervous system disorders) | 8 | 1
Difficulty Sleeping (General disorders) | 3 | 0
Eye issues (Eye disorders) | 1 | 2 — Eye strain, difficulty with night vision, and tearing issues
Dizziness (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hot flash (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT03060759/Prot_SAP_000.pdf